## Coverpage

Title: Advancement of Clinical Referral to Physical Activity for Cardiometabolic Disease

Prevention

Brief Title: The Clinical Referral to Activity Study

NCT: NCT04743856

Date Created/Modified: November 3, 2025

## Statistical Analyses

**6.1.6 Statistical Analyses**: For our primary outcomes, we hypothesize that participants randomized to ActiveGOALSv2 + PAT will have significantly larger (a) increases in step counts/day and % meeting MVPA goal of 150 minutes/week (to 12 months) compared to the active PAT control group. Descriptive analyses and graphic displays will be used to identify outliers, missing data, and pattern of attrition. To ensure rigor, the primary analytic strategy will be a linear or generalized mixed-effect models approach in which treatment group, time, and time by group interaction are treated as fixed effects, and subject is treated as a random effect to account for individual subject variability (two sided hypothesis test; .05 level). Mixed models are applicable to longitudinal datasets that contain missing observations, (assuming data is missing at random). Regression modeling will be conducted to adjust for important covariates. We will perform similar analyses to examine changes in secondary outcomes. Descriptive statistics on patient experience, beliefs/attitudes related to maintenance of PA changes, and program cost will also be reported. Mixed models are use to help account for missing data and no adjustments will be made for multiple comparisons.